CLINICAL TRIAL: NCT06626373
Title: Elderberry Consumption and Human Health: a Preliminary Investigation Into Effects on Indirect Calorimetry, Insulin Sensitivity, and Microbiome
Brief Title: Elderberry Consumption and Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18597
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Unspecified
Keywords: Obesity; Elderberry
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double (ParticipantOutcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Elderberry Juice (Experimental): Participants will consume elderberry juice twice/day for 1-week as well as our provided diet for 4 days.
  Interventions: Other: Elderberry Juice
- Placebo Comparator: Placebo beverage (Placebo Comparator): Participants will consume placebo beverage twice/day for 1-week as well as our provided diet for 4 days.
  Interventions: Other: Placebo Beverage

INTERVENTIONS:
Other: Elderberry Juice — Participants will consume elderberry juice 1-week.
  Arms: Experimental: Elderberry Juice
Other: Placebo Beverage — Participants will consume placebo beverage twice/day for 1-week.
  Arms: Placebo Comparator: Placebo beverage

SUMMARY:
The objective of this human study is to determine if the metabolic benefits observed with other anthocyanin-rich berries extend to elderberries. To accomplish this, we performed a short-term controlled feeding study in overweight but healthy volunteers in a placebo-controlled crossover clinical trial. Major study endpoints included blood glucose and insulin response to a high-carbohydrate meal challenge, indirect calorimetry, and profiling of the fecal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men between 22 and 75 years of age with a body mass index of 25 kg/m2 or above

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Have a body mass index less than 25 kg/m2
* Are younger than 22 years of age, or older than 75 years of age
* Known allergy or intolerance to elderberries
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring a special diet that is not in accord with the diet behavior requested for this study
* Adherence to restrictive (vegetarian or vegan) or extreme (fad [ex. Ketogenic or Atkins] or quick weight loss/gain) diet patterns and unwillingness to consume a conventional, omnivorous diet and maintain body weight
* Habitual use of tobacco (including vaping) products in the last 6 months
* Diagnosis or treatment of cancer in the past 3 years
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives, including blood thinning medications
* Type 2 diabetes requiring the use of medication
* Fasting blood glucose > 125 mg/dL
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Substrate oxidation | 3.5 hours
  Participants will be monitored by a metabolic cart at rest and while walking
Glucose tolerance/insulin sensitivity | 3 hours
  Blood will be collected following a meal tolerance test
Gut Microbiome analysis | 5 minutes
  Feces will be collected before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minj J, Riordan J, Teets C, Fernholz-Hartman H, Tanggono A, Lee Y, Chauvin T, Carbonero F, Solverson P. Diet-Induced Rodent Obesity Is Prevented and the Fecal Microbiome Is Improved with Elderberry (Sambucus nigra ssp. canadensis) Juice Powder. J Agric Food Chem. 2024 Jun 5;72(22):12555-12565. doi: 10.1021/acs.jafc.4c01211. Epub 2024 May 22. PMID 38776153
- [Background] Rust BM, Riordan JO, Carbonero FG, Solverson PM. One-Week Elderberry Juice Treatment Increases Carbohydrate Oxidation after a Meal Tolerance Test and Is Well Tolerated in Adults: A Randomized Controlled Pilot Study. Nutrients. 2023 Apr 25;15(9):2072. doi: 10.3390/nu15092072. PMID 37432227